CLINICAL TRIAL: NCT04739904
Title: Mechanisms of Hypoxia (in)Tolerance in Prematurely Born Individuals
Brief Title: Hypoxia Intolerance in Preterm Individuals
Acronym: PreAlti
Status: Completed | Type: Observational
Sponsor: Jozef Stefan Institute (Other)
Collaborators: University of Lausanne (Other)
Responsible Party: Principal Investigator, Tadej Debevec, Dr., Jozef Stefan Institute
Other Study IDs: PreAlti
Record Dates: First submitted 2021-01-22; First posted 2021-02-05 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Premature Birth; Hypoxia
Keywords: Acclimatization; Altitude; Preterm birth; Cardiorespiratory; Cerebrovascular; Exercise
MeSH Terms: conditions — Premature Birth; Hypoxia; Motor Activity | interventions — Sea Level Rise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm born: Premature born but otherwise healthy adults exposed to normoxic, normobaric hypoxic and hypobaric hypoxic interventions.
  Interventions: Other: Normoxia; Other: Normobaric hypoxia; Other: Hypobaric hypoxia
- Full-term control: Full-term born healthy adults exposed to normoxic, normobaric hypoxic and hypobaric hypoxic interventions.
  Interventions: Other: Normoxia; Other: Normobaric hypoxia; Other: Hypobaric hypoxia

INTERVENTIONS:
Other: Normoxia — 48 hours experimental protocol conducted at sea level
  Other Names: Normoxic condition; Sea level
Other: Normobaric hypoxia — 24 hours experimental protocol conducted in a normobaric hypoxic facility
  Other Names: Simulated altitude
Other: Hypobaric hypoxia — 72 hours experimental protocol conducted at terrestrial altitude
  Other Names: Terrestrial altitude

SUMMARY:
Reduced Hypoxic Ventilatory Response (HVR) and systemic O2 saturation subsequently leading to blunted aerobic capacity as well as decreased overall physical and cognitive performance are the main physiological challenges faced by prematurely born individuals in hypobaric hypoxia (i.e. during high altitude sojourn). While these phenomena have been described previously, the underlying mechanisms are currently unresolved. Given that the reduction in altitude-performance and its underlying mechanisms are not well understood, it is currently impossible to give evidence-based recommendation for altitude sojourns in this cohort. It is also of note, that even hypobaric hypoxia exposure during long-haul flights might be detrimental to well-being of pre-term born individuals.

The present project aims to comprehensively investigate physiological responses to altitude/hypoxia during rest and exercise in prematurely born, but otherwise healthy adults. Specifically, the investigators aim to elucidate the underlying mechanisms of the altered resting and exercise cardiovascular, respiratory, cerebral and hematological responses to hypoxia in prematurely born individuals. The obtained results from this cohort will be compared to the data from a control groups consisting of healthy, age and aerobic capacity-matched individuals born at full-term. While acute hypoxic effects will be the focus of the project's first phase, the researchers will test the effect of prolonged terrestrial (real) or simulated (normobaric hypoxia) altitude exposures in the second part. This phase will, in addition to the insight into the prolonged altitude acclimatization modulation in prematurely born individuals, also enable the potential differences between the effects of normobaric (simulated) and hypobaric (terrestrial) hypoxia in this cohort to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* prematurely born (gestational age: ≤ 32 weeks; gestational weight ≤ 1500g)
* full-term born
* healthy individuals
* male

Exclusion Criteria:

* presence of any medical risk factors to exercise and/or exposure to altitude
* presence of any medical condition that would make the protocol unreasonably hazardous for the patient
* smokers
* exposure to altitude above 1000m in the last 2 months

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Prematurely born adults involved in this study must fulfil the following characteristics at birth: gestational age ≤ 32 weeks and gestational weight ≤ 1500g.
  Conversely, full-term adults involved in this study must fulfil the following characteristics at birth: gestational age of at least 38 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Cerebrovascular reactivity to carbon dioxide (CO2) | 48 hours after exposure to normoxia and hypobaric hypoxia, respectively.
  Subjects will breath 4 min 3% CO2 and 4 min 6% CO2 separated by 4 min of breathing ambient air. Gas exchange, blood flow in the middle cerebral artery and peripheral oxygen saturation will be continuously recorded by metabolic cart, transcranial doppler, and finger pulse oximeter, respectively.
Cognitive function | 24 hours after exposure to normoxia, hypobaric hypoxia, and normobaric hypoxia, respectively
  Cognitive function will be assessed by a computerized psychometric test battery previously used by our research group. These will assess working memory and visuo-motor coordination.
Acute Mountain Sickness (AMS) | 8 hours (prior to sleep) and 16 hours (upon waking) after exposure to hypobaric and normobaric hypoxia
  AMS will be assessed by Lake Louise scale. AMS will be diagnosed if the Lake Louise score is 3 or higher.
Change in respiratory function | Immediately after exposure to hypobaric and normobaric hypoxia, relative to baseline.
  Respiratory function will be assessed by spirometry.
Lung comets | Every day before and immediately after each exercise bout.
  Lung comets will be assessed by counting the number of B-lines present, which will be measured using Doppler ultrasound.
Heart rate response to exercise | Every day before exercise, during exercise and at the instant of volitional exhaustion.
  Heart rate (HR, bpm) will be continuously monitored during different exercise bouts of variety intensities (moderate and heavy intensities will be used).
Respiratory response to exercise | Every day before exercise, during exercise and at the instant of volitional exhaustion.
  Oxygen consumption (VO2, L/min and mL/min/kg) will be continuously monitored during different exercise bouts of variety intensities (moderate and heavy intensities will be used).
Changes in muscular oxygenation during exercise | Every day before exercise, during exercise and at the instant of volitional exhaustion.
  Muscle oxygenation/deoxygenation will be continuously recorded during each exercise bout by Near Infra-Red Spectroscopy (NIRS) placed on the vastus lateralis. NIRS measure the quantity of oxygenated and deoxygenated haemoglobin and myoglobin (microM) in the investigated areas (vastus lateralis).
Changes in cerebral oxygenation during exercise | Every day before exercise, during exercise and at the instant of volitional exhaustion.
  Brain oxygenation/deoxygenation will be continuously recorded during each exercise bout by Near Infra-Red Spectroscopy (NIRS) placed at the frontal levels. NIRS measure the quantity of oxygenated and deoxygenated haemoglobin (microM) in the investigated areas (prefrontal cortex).
Changes in the rate of muscular oxygen consumption (mV̇O2) | Before each exercise bouts.
  Muscle oxygen consumption will be assessed using a previously validated protocol. Briefly, a Near Infra-Red Spectroscopy (NIRS) optode will be placed on the vastus lateralis muscle. Before the protocol, an ischemic calibration will be performed to normalize the NIRS signals by inflating the blood pressure cuff to 250-300 mmHg for a maximum of 5 min. Resting mV̇O2 will be assessed from the decrease in muscle oxygenation which accompanies the arterial occlusion. Four resting measurements will be performed using 10 sec of arterial occlusion. Then, each subject will perform a voluntary knee extension exercise for 15 sec. To measure the recovery of oxygen consumption after exercise, subject will have a series of arterial occlusion as follows: 5 occlusions 5sec on-5sec off, 5 occlusions 5sec on-5sec off, and 8 occlusions 10 sec on-20 sec off.
Acute change in sleep quality | On the first night in normoxia, normobaric hypoxia and hypobaric hypoxia.
  Polysomnography will be used to assess sleep quality. Measurements will include electroencephalography (EEG), electrooculography (EOG), chin and tibial surface electromyography (EMG), electrocardiography (ECG), nasal pressure (nasal pressure cannula), respiratory movements (chest and abdominal belts) as well as capillary oxygenated haemoglobin saturation measurement.
Change in sleep quality after prolonged exposure to hypobaric hypoxia | On the third night after exposure to terrestrial altitude.
  Polysomnography will be used to assess sleep quality. Measurements will include electroencephalography (EEG), electrooculography (EOG), chin and tibial surface electromyography (EMG), electrocardiography (ECG), nasal pressure (nasal pressure cannula), respiratory movements (chest and abdominal belts) as well as capillary oxygenated haemoglobin saturation measurement.
Changes in endothelial capacity to flow-mediated dilation (FMD) | 24 hours after exposure to normoxia and hypobaric hypoxia.
  A pneumatic cuff is positioned distal to the ultrasound probe in order to avoid ischemia of the artery studied. Radial artery diameter is measured at rest, during inflation of the distal cuff to suprasystolic pressure (5 min) and for the 5 min following deflation. The subsequent decrease in local blood flow in response to ischemia causes a progressive decrease in the radial artery diameter until a plateau (L-FMC). Upon cuff deflation, the increased blood flow causes radial artery dilatation. L-FMC is calculated as the percentage decrease in arterial diameter in the last 30 s of cuff occlusion as compared with resting diameter. FMD is calculated as the maximum percentage increase in arterial diameter following cuff deflation.
Changes in orthostatic tolerance | At 6am on every trial day (upon waking).
  Orthostatic tolerance will be assessed by measuring heart rate variability. This will involve an app-validated 10-min protocol, which will use a chest-band to monitor heart rate changes from 5 minutes of supine position followed by 5 minutes of standing.
Changes in oxidative stress markers in the blood | Blood samples will be collected at 6am (upon waking).
  Oxidative stress markers concentration will be measured on collected venous blood sample.
Change in salivary cortisol concentration | Saliva samples will be collected at 6am (upon waking).
  Cortisol concentration will be measured on collected saliva samples.
Change in hydration status | Urine samples will be collected at 6am (upon waking).
  Urine samples will be assessed using urine specific gravity.

SECONDARY OUTCOMES:
Change in cerebral blood flow in the internal carotid artery | Cerebral blood flow will be measured at 10am.
  Cerebral blood flow in the internal will be assessed every morning by doppler ultrasound.

CONTACTS AND LOCATIONS:
Locations (3):
- Slovenia (2):
  - Jozef Stefan Institute, Ljubljana
  - University of Ljubljana, Ljubljana
- Institute of Sport Sciences of the University of Lausanne, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Manferdelli G, Narang BJ, Bourdillon N, Debevec T, Millet GP. Physiological Responses to Exercise in Hypoxia in Preterm Adults: Convective and Diffusive Limitations in the O 2 Transport. Med Sci Sports Exerc. 2023 Mar 1;55(3):482-496. doi: 10.1249/MSS.0000000000003077. Epub 2022 Oct 26. PMID 36459101